CLINICAL TRIAL: NCT03150056
Title: A Phase IB Open-label, Dose Escalation and Expansion Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of GSK525762 in Combination With Androgen Deprivation Therapy and Other Agents in Subjects With Castrate-resistant Prostate Cancer (CRPC)
Brief Title: Dose Escalation and Dose Expansion Study of GSK525762 in Combination With Androgen Deprivation Therapy in Participants With Castrate-resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study has been terminated due to meeting protocol defined futility.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204697; 2016-003416-13 (EudraCT Number)
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2021-08-26 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Solid Tumours
Keywords: Abiraterone; Castrate-resistant prostate cancer; Androgen receptor targeted therapy; RP2D; Enzalutamide; GSK525762
MeSH Terms: interventions — molibresib; abiraterone; enzalutamide; Prednisone

STUDY DESIGN:
Intervention Model Description: This will be a two-arm, open-label dose escalation and dose expansion cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK525762 + Abiraterone (+ Prednisone) (Arm A) (Experimental)
  Interventions: Drug: GSK525762; Drug: Abiraterone; Drug: Prednisone
- GSK525762 + Enzalutamide (Arm B) (Experimental)
  Interventions: Drug: GSK525762; Drug: Enzalutamide

INTERVENTIONS:
Drug: GSK525762 — GSK525762 will be administered.
Drug: Abiraterone — Abiraterone will be administered.
  Arms: GSK525762 + Abiraterone (+ Prednisone) (Arm A)
Drug: Enzalutamide — Enzalutamide will be administered.
  Arms: GSK525762 + Enzalutamide (Arm B)
Drug: Prednisone — Prednisone will be administered as a concomitant medication in combination with abiraterone
  Arms: GSK525762 + Abiraterone (+ Prednisone) (Arm A)

SUMMARY:
This study aims to evaluate the combination of GSK525762 with other agents that have been shown to be effective in the treatment of CRPC or metastatic (m)CRPC. This study is designed to determine the maximum tolerated dose (MTD) and recommended Phase II dose (RP2D) based on safety, tolerability, pharmacokinetic, and efficacy profiles of GSK525762 in combination with either abiraterone (Arm A) or enzalutamide (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Males >=18 years of age (at the time written consent is obtained for screening).
* Histologically confirmed adenocarcinoma of the prostate: screening and on-treatment biopsy is mandatory. If adequate number of paired biopsy samples are collected (>=20 paired samples for each dose level in each Arm, unless an Arm is closed early), then further biopsy sampling will be considered based on available data; screening biopsy can be waived if participant had a recent biopsy after failure of the most recent therapy (within 30 days) and the biopsy sample is secured to be sent as screening biopsy for this study.
* Surgically or medically castrated, with testosterone levels of less than or equal to (<=)50 nanograms per deciliter (ng/dL) (<2.0 nanometer [nM]). If the participant is being treated with luteinizing hormone-releasing hormone (LHRH) agonists/antagonists (participant who have not undergone orchiectomy) this therapy must have been initiated at least 4 weeks prior to Week 1 Day 1 and must be continued throughout the study.
* Participants must have failed prior therapy with abiraterone, enzalutamide, or both:

  1. Has completed at least 12 weeks of prior continuous therapy with abiraterone or enzalutamide in any prior line.
  2. Lead-in dosing period for enzalutamide only will be required under the following circumstance:

  (i) If the participant has enzalutamide discontinuation for >7 days prior to dosing start with GSK525762 plus enzalutamide on trial, then a enzalutamide only lead-in dosing of 28 days is required.

(ii) If the participant has enzalutamide discontinuation for <=7 days prior to dosing start with GSK525762 plus enzalutamide on trial, then an enzalutamide only lead-in dosing of 14 days is required.

(iii) If the participant is on continuous dosing with enzalutamide prior to dosing start with GSK525762 plus enzalutamide on trial, then participant can start on combined dosing at end of screening period.

(c) Lead-in dosing period for abiraterone only will be required: if the participant has abiraterone discontinuation for more than 3 days prior to dosing start with GSK525762 plus abiraterone on trial, then abiraterone only lead-in dosing of 7 days is required.

* One to two line(s) of prior taxane-based chemotherapy allowed. If docetaxel chemotherapy is used more than once, this will be considered as one regimen. Participants who have not received prior chemotherapy in any setting will qualify for study if they are ineligible for or refuse chemotherapy.
* Documented prostate cancer progression as assessed by the investigator with one of the following:

  1. PSA progression defined by a minimum of 3 rising PSA levels with an interval of >=1 week between each determination. The PSA value at screening must be >=5 microgram (µg)/Liter (L) (5 ng/mL) if PSA is the only indication of progression; participants on systemic glucocorticoids for control of symptoms must have documented PSA progression by PCWG3 while on systemic glucocorticoids prior to commencing Week 1 Day 1 treatment.
  2. Radiographic progression of soft tissue disease by PCWG3-modified RECIST 1.1 criteria or bone metastasis with 2 or more documented new bone lesions on a bone scan with or without PSA progression.
* ECOG performance status of 0 or 1.
* Life expectancy >12 weeks.
* Able to swallow and retain orally administered medication.
* Must have adequate organ function.
* Male participants are eligible to participate if they agree to use contraceptive methods.

Exclusion Criteria:

* Surgery or local prostatic intervention (excluding a prostatic biopsy) less than 28 days of Week 1 Day 1.
* Participants with neuroendocrine and/or small cell CRPC.
* Recent prior therapy, defined as:

  1. Any investigational or approved non-biologic anti-cancer drug within 14 days prior to the first dose of GSK525762 and abiraterone/enzalutamide.
  2. Any nitrosoureas or mitomycin C within 42 days prior to the first dose of GSK525762 and abiraterone/enzalutamide.
  3. Any anti-cancer biologic agents within five half-lives prior to the first dose of GSK525762 and abiraterone/enzalutamide.
  4. If the participant received radiotherapy <90 days prior to study treatment, the irradiated lesion cannot be the only lesion used for evaluating response.
  5. Any major surgery within 28 days prior to the first dose of GSK525762 and abiraterone/enzalutamide.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, cardiac disease, or clinically significant bleeding episodes). Any serious and/or unstable pre-existing medical (aside from malignancy), psychiatric disorder, or other conditions that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator; systolic blood pressure higher than 150 millimeter of mercury (mmHg) or diastolic blood pressure higher than 90 mmHg found on 2 separate occasions separated by 1 week, despite adequate therapy, will be defined as uncontrolled hypertension; uncontrolled diabetes mellitus (despite therapeutic, compliance intervention) as defined by a hemoglobin A1c (HbA1c) level more than 8% and/or occurrence of more than 2 episodes of ketoacidosis in the 12 months prior to the first dose of study drug.
* Cardiac abnormalities as evidenced by any of the following:

  1. Baseline QT interval corrected for heart rate by Fridericia's formula (QTcF) interval >=480 milliseconds (msec).
  2. Clinically significant conduction abnormalities or arrhythmias, such as participants with second degree (Type II) or third degree atrio-ventricular block.
  3. History or evidence of current >=Class II congestive heart failure as defined by New York Heart Association (NYHA).
  4. History of acute coronary syndromes (including unstable angina and myocardial infarction), coronary angioplasty, or stenting within the past 3 months. Participants with a history of stent placement requiring ongoing anti-coagulant therapy (e.g., clopidogrel, prasugrel) will not be permitted to enroll.
  5. Known cardiac metastasis.
* Participants with history of known bleeding disorder(s) or history of clinically significant hemorrhage (e.g., gastrointestinal, neurologic), within the past 6 months.
* Therapeutic-dose anticoagulation (e.g., warfarin, low-molecular weight heparin [LMWH], or novel oral anticoagulants) must be discontinued and coagulation parameters must be normalized prior to the first dose of GSK525762 and abiraterone/enzalutimide. Prophylactic anticoagulation, with low doses (per standard practice) of agents such as LMWH, direct thrombin inhibitors, or factor Xa inhibitors is permitted.
* Concurrent use of high dose aspirin (doses up to 81 milligrams (mg) oral dose daily allowed, or 100 mg, as per country standards) and non-steroidal anti-inflammatory drugs (NSAIDS), except for where NSAIDs provide documented benefit over other analgesics, and then to be used with caution including concomitant use of proton pump inhibitors).
* Any acute toxicities due to prior chemotherapy and / or radiotherapy that have not resolved to a National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 grade <=1 with the exception of chemotherapy induced alopecia and grade 2 peripheral neuropathy.
* The participant has an active second malignancy other than curatively resected basal cell or squamous cell carcinoma of the skin, in situ carcinoma of the bladder, or other cancers for which they are treated with curative intent with no active disease in the 3 years prior to enrollment.
* Participants with known symptomatic brain metastasis are not suitable for enrolment. Participants with asymptomatic, stable, treated brain metastases are eligible for study entry.
* History of seizure within 6 months of study treatment initiation or any condition that may predispose participant to seizure (e.g., prior cortical stroke or significant brain trauma) or who are currently being treated with cytochrome P450 enzyme inducing anti-epileptic drugs for seizures (use of anti-epileptic drugs to control pain is allowed in participants not suffering from seizures unless drug is excluded due to Cytochrome (CY)P3A4 induction - phenytoin, carbamazepine, phenobarbital).
* History of loss of consciousness or transient ischemic attack within 12 months prior to enrollment.
* Participants with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable and asymptomatic.
* Current use of a prohibited medication or planned use of any forbidden medications during treatment with GSK525762 and abiraterone/enzalutamide. This includes medications that are potent inducers or inhibitors of CYP3A4 enzymes or strong inhibitors of CYP2C8.
* Participants with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Participants with known bleeding diathesis.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment).
* Initiating bisphosphonate or denosumab therapy or adjusting dose/regimen within 3 months prior to Week 1 Day 1. Participants on a stable bisphosphonate or denosumab therapy are eligible and may continue.
* Any serious known immediate or delayed hypersensitivity reaction to GSK525762 or idiosyncrasy to drugs chemically related to the investigational drugs. Additionally, any known hypersensitivity to either enzalutamide, abiraterone or any excipients would be excluded.
* Known history of human immunodeficiency virus (HIV).
* Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 73 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- United States (9):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Madison, Wisconsin
- Australia (3):
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Santander
- United Kingdom (2):
  - GSK Investigational Site, Sutton, London
  - GSK Investigational Site, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, dose escalation and expansion study to investigate safety, pharmacokinetics, pharmacodynamics and clinical activity of GSK525762 in combination with abiraterone or enzalutamide in participants with castrate resistant prostate cancer (CRPC).
Pre-assignment Details: This study has been terminated due to meeting protocol defined futility. A total of 73 participants were enrolled in the study.
Groups:
- GSK525762 60 mg+Abiraterone 1000 mg: Participants received once daily oral dose of GSK525762 60 milligram (mg) in combination with abiraterone 1000 mg up to maximum of 21.3 months. Participants received prednisone 5 mg orally twice daily as per abiraterone label.
- GSK525762 60 mg Alternate+Abiraterone 1000 mg: Participants received an alternate dosing schedule- once daily GSK525762 60 mg + abiraterone 1000 mg tablets via the oral route for 2 weeks followed by 1 week off-treatment up to maximum of 21.3 months. Participants received prednisone 5 mg orally twice daily as per abiraterone label.
- GSK525762 40 mg+Abiraterone 1000 mg: Participants received once daily oral dose of GSK525762 40 mg in combination with abiraterone 1000 mg up to maximum of 21.3 months. Participants received prednisone 5 mg orally twice daily as per abiraterone label.
- GSK525762 80 mg+Enzalutamide 160 mg: Participants received once daily oral dose of GSK525762 80 mg in combination with enzalutamide 160 mg up to maximum of 21.3 months.
- GSK525762 60 mg+Enzalutamide 160 mg: Participants received once daily oral dose of GSK525762 60 mg in combination with enzalutamide 160 mg up to maximum of 21.3 months.
- GSK525762 60 mg Alternate+Enzalutamide 160 mg: Participants received an alternate dosing schedule- once daily GSK525762 60 mg + enzalutamide 160 mg tablets via the oral route for 2 weeks followed by 1 week off-treatment up to maximum of 21.3 months.
Period: Overall Study
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Started | 10 | 6 | 4 | 10 | 22 | 21
Completed | 0 | 1 | 1 | 2 | 9 | 3
Not Completed | 10 | 5 | 3 | 8 | 13 | 18
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Study terminated by Sponsor | 1 | 3 | 1 | 1 | 5 | 6
Not completed — Death | 9 | 2 | 2 | 7 | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg | Total
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21 | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.4 (7.69) | 68.0 (9.57) | 76.3 (4.11) | 69.3 (4.72) | 71.0 (6.49) | 69.1 (5.11) | 70.2 (6.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 6 | 4 | 10 | 22 | 21 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-East Asian Heritage | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 1 | 0 | 0 | 0 | 1 | 1 | 3
  White-Arabic/North African Heritage | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White-White/Caucasian/European Heritage | 7 | 6 | 4 | 10 | 21 | 19 | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, any other situation according to medical or scientific judgement, or is associated with liver injury and impaired liver function.
Time Frame: Up to 21.3 months
Population: All Treated Population consisted of all participants who received at least one dose of GSK525762 or abiraterone or enzalutamide.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21
Participants
  Any AEs | 10 | 6 | 4 | 10 | 22 | 21
  Any SAEs | 4 | 2 | 0 | 1 | 6 | 7

2. Primary Outcome: Number of Participants With AEs Leading to Any Dose Reduction or Delays
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with AEs leading to any dose reduction or delays have been presented.
Time Frame: Up to 21.3 months
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21
Participants
  Dose reduction | 4 | 1 | 0 | 7 | 10 | 7
  Dose delay | 5 | 2 | 4 | 8 | 15 | 12

3. Primary Outcome: Number of Participants Who Withdrew Due to Toxicity and Changes in Safety Assessment
Description: Number of participants who withdrew due to toxicity and changes in safety assessment including laboratory parameters and vital signs have been presented.
Time Frame: Up to 21.3 months
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21
Participants | 6 | 2 | 2 | 3 | 8 | 4

4. Primary Outcome: Percentage of Participants With Greater Than or Equals to (>=)50 Percent (%) Decrease in Prostate-specific Antigen From Baseline (PSA50)
Description: PSA50 response rate is defined as percentage of participants with a decrease of >=50% in the PSA concentration from the Baseline PSA value determined at least 12 weeks after start of treatment and confirmed >=4 weeks later by an additional PSA evaluation.
Time Frame: Up to 21.3 months
Population: Modified All Treated Population comprised of all participants who received at least one dose of GSK525762 plus abiraterone/enzalutamide. Only those participants with data available at the indicated time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 19 | 21
Percentage of participants | 0 [0.0 to 30.8] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 0 [0.0 to 30.8] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1]

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK525762 and Its Active Metabolites GSK3529246
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK525762 and GSK3529246 (metabolite of GSK525762). PK parameters were calculated using standard non-compartmental analysis. PK Population consisted of all participants from the All Treated Safety Population for whom a PK sample was obtained and analyzed.
Time Frame: Pre-dose, 30 minutes, 1, 3, 6 to 12, 24 hours post-dose on Day 1 of Weeks 1 and 3
Population: PK Population. Only those participants with data available at the indicated time points were analyzed (indicated by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 21 | 18
Nanogram per milliliter
  GSK525762:Week1 Day1,n=10,6,4,10,21,18 | 950.319 (19.18) | 993.154 (33.77) | 671.129 (30.44) | 427.580 (31.76) | 333.256 (48.86) | 336.296 (43.28)
  GSK525762:Week3 Day1,n=4,3,3,9,17,10: number analyzed (Participants) | 4 | 3 | 3 | 9 | 17 | 10
  GSK525762:Week3 Day1,n=4,3,3,9,17,10 | 891.302 (36.79) | 735.171 (21.63) | 559.711 (40.59) | 284.298 (45.12) | 158.409 (153.45) | 171.527 (47.88)
  GSK3529246:Week1 Day1,n=10,6,4,10,21,18 | 280.892 (43.14) | 318.772 (31.13) | 199.456 (32.94) | 408.208 (39.86) | 321.750 (24.24) | 323.685 (25.77)
  GSK3529246:Week3 Day1,n=4,3,3,10,17,10: number analyzed (Participants) | 4 | 3 | 3 | 10 | 17 | 10
  GSK3529246:Week3 Day1,n=4,3,3,10,17,10 | 447.929 (39.30) | 444.232 (26.74) | 364.151 (15.46) | 449.614 (49.54) | 328.398 (39.74) | 356.615 (18.26)

6. Secondary Outcome: Time to Cmax (Tmax) of GSK525762 and Its Active Metabolites GSK3529246
Description: Blood samples were collected at indicated time points for PK analysis of GSK525762 and GSK3529246 (metabolite of GSK525762). PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 30 minutes, 1, 3, 6 to 12, 24 hours post-dose on Day 1 of Weeks 1 and 3
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 21 | 18
Hours
  GSK525762:Week1 Day1,n=10,6,4,10,21,18 | 0.800 [0.50 to 2.92] | 0.558 [0.50 to 1.00] | 1.000 [0.58 to 3.08] | 0.508 [0.40 to 1.08] | 1.000 [0.45 to 3.00] | 0.742 [0.50 to 6.00]
  GSK525762:Week3 Day1,n=4,3,3,9,17,10: number analyzed (Participants) | 4 | 3 | 3 | 9 | 17 | 10
  GSK525762:Week3 Day1,n=4,3,3,9,17,10 | 0.500 [0.50 to 0.50] | 1.000 [0.50 to 3.00] | 0.950 [0.50 to 1.00] | 0.583 [0.47 to 3.00] | 0.933 [0.00 to 3.03] | 0.517 [0.50 to 3.08]
  GSK3529246:Week1 Day1,n=10,6,4,10,21,18 | 3.000 [1.18 to 6.00] | 3.000 [0.53 to 6.00] | 2.042 [1.00 to 3.08] | 2.067 [1.00 to 3.00] | 2.917 [0.53 to 6.05] | 1.817 [0.95 to 6.00]
  GSK3529246:Week3 Day1,n=4,3,3,10,17,10: number analyzed (Participants) | 4 | 3 | 3 | 10 | 17 | 10
  GSK3529246:Week3 Day1,n=4,3,3,10,17,10 | 1.000 [0.85 to 3.00] | 3.000 [1.00 to 6.17] | 3.000 [1.00 to 3.03] | 1.042 [0.50 to 6.00] | 1.017 [0.00 to 6.00] | 1.875 [0.50 to 6.33]

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval (AUC[0-tau]) of GSK525762 and Its Active Metabolites GSK3529246
Description: as for outcome 6
Time Frame: Pre-dose, 30 minutes, 1, 3, 6 to 12, 24 hours post-dose on Day 1 of Weeks 1 and 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 8 | 2 | 3 | 6 | 12 | 10
Hours*nanogram per milliliter
  GSK525762:Week1 Day1,n=8,2,2,6,9,8: number analyzed (Participants) | 8 | 2 | 2 | 6 | 9 | 8
  GSK525762:Week1 Day1,n=8,2,2,6,9,8 | 4927.834 (71.78) | 4677.411 (21.59) | 4172.282 (31.08) | 1139.481 (34.32) | 1261.529 (102.14) | 959.452 (60.97)
  GSK525762:Week3 Day1,n=4,1,3,5,6,6: number analyzed (Participants) | 4 | 1 | 3 | 5 | 6 | 6
  GSK525762:Week3 Day1,n=4,1,3,5,6,6 | 2697.923 (69.10) | 2580.877 (NA) — Geometric coefficient of variation could not be calculated for a single participant. | 1561.908 (13.67) | 674.437 (57.10) | 660.607 (14.41) | 386.950 (37.03)
  GSK3529246:Week1 Day1,n=2,1,0,5,9,10: number analyzed (Participants) | 2 | 1 | 0 | 5 | 9 | 10
  GSK3529246:Week1 Day1,n=2,1,0,5,9,10 | 3765.196 (0.47) | 4918.549 (NA) — Geometric coefficient of variation could not be calculated for a single participant. |  | 4379.342 (30.76) | 3373.990 (19.73) | 3306.018 (31.84)
  GSK3529246:Week3 Day1,n=2,2,2,4,12,7: number analyzed (Participants) | 2 | 2 | 2 | 4 | 12 | 7
  GSK3529246:Week3 Day1,n=2,2,2,4,12,7 | 4170.516 (6.55) | 5146.749 (9.99) | 4598.235 (16.28) | 3816.407 (37.02) | 3386.702 (30.44) | 3082.516 (33.36)

8. Secondary Outcome: Trough Concentration (Ctrough) of GSK525762 and Its Active Metabolites GSK3529246
Description: as for outcome 6
Time Frame: Pre-dose, 30 minutes, 1, 3, 6 to 12, 24 hours post-dose on Day 1 of Weeks 1 and 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 8 | 3 | 3 | 9 | 20 | 17
Nanogram per milliliter
  GSK525762:Week1 Day1,n=8,2,3,1,3,4: number analyzed (Participants) | 8 | 2 | 3 | 1 | 3 | 4
  GSK525762:Week1 Day1,n=8,2,3,1,3,4 | 22.418 (192.37) | 8.696 (72.93) | 13.664 (119.83) | 2.100 (NA) — Geometric coefficient of variation could not be calculated for a single participant. | 5.053 (3035.92) | 1.660 (34.60)
  GSK525762:Week3 Day1,n=2,2,2,1,0,0: number analyzed (Participants) | 2 | 2 | 2 | 1 | 0 | 0
  GSK525762:Week3 Day1,n=2,2,2,1,0,0 | 8.966 (93.46) | 4.555 (522.90) | 1.410 (48.34) | 3.540 (NA) — Geometric coefficient of variation could not be calculated for a single participant. |  |
  GSK3529246:Week1 Day1,n=8,3,3,9,20,17 | 58.995 (52.50) | 68.379 (47.51) | 42.107 (52.26) | 46.011 (38.73) | 37.765 (56.41) | 38.200 (53.15)
  GSK3529246:Week3 Day1,n=3,3,2,7,13,8: number analyzed (Participants) | 3 | 3 | 2 | 7 | 13 | 8
  GSK3529246:Week3 Day1,n=3,3,2,7,13,8 | 48.223 (99.09) | 48.291 (29.86) | 63.526 (3.90) | 50.882 (77.10) | 32.299 (60.18) | 26.165 (76.95)

9. Secondary Outcome: Cmax of Abiraterone
Description: Blood samples were collected at indicated time points for PK analysis of abiraterone. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 30 minutes, 1, 3, 6 to 12, 24 hours post-dose on Day 1 of Weeks 1 and 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg
Number analyzed (Participants) | 10 | 5 | 4
Nanogram per milliliter
  Week 1 Day 1, n=10,5,4 | 77.962 (57.07) | 63.369 (114.31) | 122.496 (131.30)
  Week 3 Day 1, n=4,4,2: number analyzed (Participants) | 4 | 4 | 2
  Week 3 Day 1, n=4,4,2 | 149.673 (65.39) | 87.554 (110.92) | 146.924 (76.98)

10. Secondary Outcome: Tmax of Abiraterone
Description: as for outcome 9
Time Frame: Pre-dose, 30 minutes, 1, 3, 6 to 12, 24 hours post-dose on Day 1 of Weeks 1 and 3
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg
Number analyzed (Participants) | 10 | 5 | 4
Hours
  Week 1 Day 1, n=10,5,4 | 1.133 [0.17 to 3.13] | 1.083 [0.53 to 3.00] | 0.750 [0.00 to 1.08]
  Week 3 Day 1, n=4,4,2: number analyzed (Participants) | 4 | 4 | 2
  Week 3 Day 1, n=4,4,2 | 1.000 [0.85 to 1.00] | 2.000 [0.98 to 3.00] | 3.017 [3.00 to 3.03]

11. Secondary Outcome: AUC(0-tau) of Abiraterone
Description: as for outcome 9
Time Frame: Pre-dose, 30 minutes, 1, 3, 6 to 12, 24 hours post-dose on Day 1 of Weeks 1 and 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg
Number analyzed (Participants) | 5 | 2 | 1
Hours*nanogram per milliliter
  Week 1 Day 1, n=5,1,1: number analyzed (Participants) | 5 | 1 | 1
  Week 1 Day 1, n=5,1,1 | 432.368 (56.74) | 148.871 (NA) — Geometric coefficient of variation could not be calculated for a single participant. | 1405.809 (NA) — Geometric coefficient of variation could not be calculated for a single participant.
  Week 3 Day 1, n=1,2,1: number analyzed (Participants) | 1 | 2 | 1
  Week 3 Day 1, n=1,2,1 | 1361.627 (NA) — Geometric coefficient of variation could not be calculated for a single participant. | 595.686 (64.72) | 2185.039 (NA) — Geometric coefficient of variation could not be calculated for a single participant.

12. Secondary Outcome: Ctrough of Abiraterone
Description: as for outcome 9
Time Frame: Pre-dose, 30 minutes, 1, 3, 6 to 12, 24 hours post-dose on Day 1 of Weeks 1 and 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg
Number analyzed (Participants) | 9 | 4 | 3
Nanogram per milliliter
  Week 1 Day 1, n=9,2,3: number analyzed (Participants) | 9 | 2 | 3
  Week 1 Day 1, n=9,2,3 | 7.603 (93.00) | 4.636 (1802.64) | 11.263 (86.21)
  Week 3 Day 1, n=2,4,1: number analyzed (Participants) | 2 | 4 | 1
  Week 3 Day 1, n=2,4,1 | 15.114 (9.84) | 7.697 (69.99) | 21.800 (NA) — Geometric coefficient of variation could not be calculated for a single participant.

13. Secondary Outcome: Cmax of Enzalutamide
Description: Blood samples were collected at indicated time points for PK analysis of enzalutamide. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose on Day 1 of Weeks 1, 3, 5, 9, 17 and 25
Population: PK Population. Cmax could not be derived as only pre-dose samples were collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 22 | 21
Microgram per milliliter | NA (NA) — Cmax could not be derived as only pre-dose samples were collected. | NA (NA) — Cmax could not be derived as only pre-dose samples were collected. | NA (NA) — Cmax could not be derived as only pre-dose samples were collected.

14. Secondary Outcome: Tmax of Enzalutamide
Description: as for outcome 13
Time Frame: Pre-dose on Day 1 of Weeks 1, 3, 5, 9, 17 and 25
Population: PK Population. Tmax could not be derived as only pre-dose samples were collected.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 22 | 21
Hours | NA [NA to NA] — Tmax could not be derived as only pre-dose samples were collected. | NA [NA to NA] — Tmax could not be derived as only pre-dose samples were collected. | NA [NA to NA] — Tmax could not be derived as only pre-dose samples were collected.

15. Secondary Outcome: AUC(0-tau) of Enzalutamide
Description: as for outcome 13
Time Frame: Pre-dose on Day 1 of Weeks 1, 3, 5, 9, 17 and 25
Population: PK Population. AUC(0-tau) could not be derived as only pre-dose samples were collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 22 | 21
Hours*microgram per milliliter | NA (NA) — AUC(0-tau) could not be derived as only pre-dose samples were collected | NA (NA) — AUC(0-tau) could not be derived as only pre-dose samples were collected | NA (NA) — AUC(0-tau) could not be derived as only pre-dose samples were collected

16. Secondary Outcome: Ctrough of Enzalutamide
Description: as for outcome 13
Time Frame: Pre-dose on Day 1 of Weeks 1, 3, 5, 9, 17 and 25
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 20 | 18
Microgram per milliliter
  Week 1 Day 1, Pre-dose, n=9,20,18: number analyzed (Participants) | 9 | 20 | 18
  Week 1 Day 1, Pre-dose, n=9,20,18 | 13.066 (21.74) | 13.313 (21.70) | 14.546 (30.34)
  Week 3 Day 1, Pre-dose, n=9,19,13: number analyzed (Participants) | 9 | 19 | 13
  Week 3 Day 1, Pre-dose, n=9,19,13 | 10.385 (23.30) | 10.902 (24.96) | 11.497 (27.34)
  Week 5 Day 1, Pre-dose, n=10,15,18: number analyzed (Participants) | 10 | 15 | 18
  Week 5 Day 1, Pre-dose, n=10,15,18 | 10.026 (21.80) | 9.814 (44.21) | 12.561 (31.27)
  Week 9 Day 1, Pre-dose, n=6,6,13: number analyzed (Participants) | 6 | 6 | 13
  Week 9 Day 1, Pre-dose, n=6,6,13 | 10.021 (27.01) | 8.064 (85.90) | 12.056 (30.12)
  Week 17 Day 1, Pre-dose, n=4,2,4: number analyzed (Participants) | 4 | 2 | 4
  Week 17 Day 1, Pre-dose, n=4,2,4 | 8.621 (22.86) | 12.568 (10.14) | 10.267 (58.45)
  Week 25 Day 1, Pre-dose, n=2,2,2: number analyzed (Participants) | 2 | 2 | 2
  Week 25 Day 1, Pre-dose, n=2,2,2 | 10.103 (8.13) | 13.069 (9.75) | 13.791 (5.13)

17. Secondary Outcome: Disease Control Rate at Week 24
Description: Disease control rate (DCR) is defined as the percentage of participants with >=1 post-Baseline disease assessment who showed either a confirmed complete response (CR), partial response (PR) or stable disease (SD) observed at >=24 weeks per prostate cancer working group 3 (PCWG3)-modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1; where CR: disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeter in the short axis; PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive diseases. Confidence interval (CI) was computed using exact two sided 95% CI.
Time Frame: Week 24
Population: Modified All Treated Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 9 | 5 | 4 | 10 | 19 | 21
Percentage of participants | 0 [0.0 to 33.6] | 40 [5.3 to 85.3] | 50 [6.8 to 93.2] | 40 [12.2 to 73.8] | 11 [1.3 to 33.1] | 29 [11.3 to 52.2]

18. Secondary Outcome: Composite Response Rate
Description: Composite response rate was defined as the percentage of participants with one of the following: a) Response based on PCWG3-modified RECIST version 1.1, b) PSA decrease of >=50% from Baseline at Week 12 and thereafter, or c) Circulating Tumor-cell Count Conversion from unfavorable (>=5/7.5 milliliter [mL]) at Baseline to favorable (<5/7.5 mL) confirmed by a second assessment at least 4 weeks later. If a participant met at least one of the above requirements, then that participant was considered a composite responder. CI was computed using exact two sided 95% CI.
Time Frame: Up to 21.3 months
Population: Modified All Treated Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21
Percentage of participants | 0 [0.0 to 30.8] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 10 [0.3 to 44.5] | 5 [0.1 to 22.8] | 0 [0.0 to 16.1]

19. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) is defined as the percentage of participants with a confirmed CR or PR at any time as per PCWG3-modified RECIST version 1.1; where CR: Disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeter (mm) in the short axis and PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters.
Time Frame: Up to 21.3 months
Population: Modified All Treated Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 9 | 5 | 4 | 10 | 19 | 21
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Circulating Tumor Cells (CTC) Response Rate
Description: CTC response rate is defined as the percentage of participants with a CTC conversion to <5/7.5 mL blood at nadir (confirmed by a second consecutive value obtained four or more weeks later) for participants with unfavourable CTC (>=5/7.5 mL) at Baseline. CI was computed using exact two sided 95% CI.
Time Frame: Up to 21.3 months
Population: Modified All Treated Population. Only those participants with data available at the indicated time points were analyzed. For GSK525762 40 mg+Abiraterone 1000 mg arm, there were no unfavorable values at Baseline, hence CTC response rate (change from unfavorable to favorable) could not be derived for this arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 7 | 3 | 0 | 3 | 12 | 11
Percentage of participants | 0 [0.0 to 41.0] | 0 [0.0 to 70.8] |  | 33 [0.8 to 90.6] | 8 [0.2 to 38.5] | 0 [0.0 to 28.5]

21. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate at Week 4
Description: PSA Response Rate is defined as percentage of participants achieving >=30% decrease from Baseline PSA after 4 weeks of study treatment. The CI was calculated using exact two sided 95% CI for the percentage of participants with Baseline PSA values who show >=30% reduction in PSA at >=4 weeks post-Baseline.
Time Frame: Week 4
Population: Modified All Treated Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21
Percentage of participants | 0 [0.0 to 30.8] | 17 [0.4 to 64.1] | 0 [0.0 to 60.2] | 0 [0.0 to 30.8] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1]

22. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from date of first dose of study treatment to date of disease progression defined as one or more of the following criteria: 1. Radiographic progression by PCWG3-modified RECIST version 1.1 for participants with measurable disease, 2. Bone progression on bone scan according to the PCGW3 criteria, 3. PSA progression according to the PCWG3 criteria accompanied by any one of the following: investigator-defined clinical progression or either of the above RECIST version 1.1 radiographic progression or bone progression.
Time Frame: Up to 21.3 months
Population: Modified All Treated Population.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21
Days | 88.0 [36.0 to 88.0] | NA [86.0 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived. | NA [36.0 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived. | 87.0 [85.0 to 112.0] | 86.0 [56.0 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 84.0 [52.0 to 330.0]

23. Secondary Outcome: Radiographic Progression-free Survival (rPFS)
Description: rPFS is defined as the time from study treatment start until the first date of either disease progression or death due to any cause. The date of disease progression is defined as the earliest date of disease progression as assessed by the investigator using PCWG3-modified RECIST, version 1.1 or progression on bone scan. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started.
Time Frame: Up to 21.3 montths
Population: Modified All Treated Population.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21
Days | 53.0 [29.5 to 165.0] | NA [NA to NA] — <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived. | NA [36.0 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived. | 416.0 [165.0 to 421.0] | 141.0 [56.0 to 220.0] | 330.0 [52.0 to 333.0]

24. Secondary Outcome: Number of Participants With Worst-Case Post Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Performance status assessments were based on 6-point ECOG scale (from 0 to 5), where 0=fully active, able to carry on all pre-disease performance without restriction; 1=restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light house work, office work); 2=ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3=capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed or chair; and 5=dead. Data for worst case post-Baseline is presented.
Time Frame: Up to 21.3 months
Population: All Treated Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 21 | 21
Participants
  0 | 2 | 0 | 0 | 2 | 1 | 1
  1 | 7 | 4 | 3 | 5 | 16 | 13
  2 | 1 | 2 | 0 | 3 | 3 | 6
  3 | 0 | 0 | 1 | 0 | 1 | 1
  4 | 0 | 0 | 0 | 0 | 0 | 0
  5 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30): Global Health Status (GHS)
Description: EORTC QLQ-C30 includes 30-items with single and multi-item scales. These included 5 functional scales (physical functioning, role functioning, cognitive functioning, emotional functioning and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a GHS/ Quality-of-Life (QoL) scale, and six single items (constipation, diarrhea, insomnia, dyspnea, appetite loss and financial difficulties). Response options for GHS/QoL range from 1 to 4, where 1=not at all and 4=very much. Scores were averaged and transformed to a 0 to 100 scale, with higher scores representing a high QoL. Baseline is defined as the latest non-missing assessment time-point prior to the first study treatment dose. Change from Baseline was calculated as post-Baseline visit value minus Baseline value.
Time Frame: Baseline (Week 1 Day 1, pre-dose) and on Day 1 of Weeks 1, 2, 3, 4, 5, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 61
Population: Modified All Treated Population. Only those participants with data available at the indicated time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 6 | 1 | 2 | 4 | 6 | 10
Scores on a scale
  Week 1 Day 1,n=1,0,0,0,2,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 0
  Week 1 Day 1,n=1,0,0,0,2,0 | 8.3 (NA) — Standard deviation could not be calculated for single participant. |  |  |  | 4.2 (5.89) |
  Week 2 Day 1,n=6,1,2,4,4,8: number analyzed (Participants) | 6 | 1 | 2 | 4 | 4 | 8
  Week 2 Day 1,n=6,1,2,4,4,8 | -8.3 (12.91) | 16.7 (NA) — Standard deviation could not be calculated for single participant. | -12.5 (29.46) | -2.1 (4.17) | 0.0 (13.61) | -1.0 (12.94)
  Week 3 Day 1,n=6,0,1,4,3,7: number analyzed (Participants) | 6 | 0 | 1 | 4 | 3 | 7
  Week 3 Day 1,n=6,0,1,4,3,7 | -8.3 (23.57) |  | -16.7 (NA) — Standard deviation could not be calculated for single participant. | -4.2 (8.33) | 2.8 (4.81) | -1.2 (3.15)
  Week 4 Day 1,n=6,1,2,3,6,10: number analyzed (Participants) | 6 | 1 | 2 | 3 | 6 | 10
  Week 4 Day 1,n=6,1,2,3,6,10 | -8.3 (10.54) | 16.7 (NA) — Standard deviation could not be calculated for single participant. | 0.0 (11.79) | 5.6 (9.62) | 1.4 (9.74) | 2.5 (16.22)
  Week 5 Day 1,n=3,0,1,3,5,9: number analyzed (Participants) | 3 | 0 | 1 | 3 | 5 | 9
  Week 5 Day 1,n=3,0,1,3,5,9 | -8.3 (14.43) |  | 8.3 (NA) — Standard deviation could not be calculated for single participant. | -5.6 (9.62) | 0.0 (11.79) | -0.0 (11.02)
  Week 9 Day 1,n=2,0,1,2,3,6: number analyzed (Participants) | 2 | 0 | 1 | 2 | 3 | 6
  Week 9 Day 1,n=2,0,1,2,3,6 | -12.5 (17.68) |  | -8.3 (NA) — Standard deviation could not be calculated for single participant. | -20.8 (5.89) | -30.6 (12.73) | -12.5 (10.21)
  Week 13 Day 1,n=1,1,1,1,2,3: number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3
  Week 13 Day 1,n=1,1,1,1,2,3 | -25.0 (NA) — Standard deviation could not be calculated for single participant. | 8.3 (NA) — Standard deviation could not be calculated for single participant. | 0.0 (NA) — Standard deviation could not be calculated for single participant. | 0.0 (NA) — Standard deviation could not be calculated for single participant. | -8.3 (11.79) | 0.0 (0.00)
  Week 17 Day 1,n=1,1,1,1,1,3: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 3
  Week 17 Day 1,n=1,1,1,1,1,3 | -25.0 (NA) — Standard deviation could not be calculated for single participant. | -16.7 (NA) — Standard deviation could not be calculated for single participant. | 16.7 (NA) — Standard deviation could not be calculated for single participant. | 0.0 (NA) — Standard deviation could not be calculated for single participant. | 0.0 (NA) — Standard deviation could not be calculated for single participant. | -11.1 (19.25)
  Week 21 Day 1,n=0,0,1,1,0,2: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 2
  Week 21 Day 1,n=0,0,1,1,0,2 |  |  | 16.7 (NA) — Standard deviation could not be calculated for single participant. | 0.0 (NA) — Standard deviation could not be calculated for single participant. |  | -4.2 (5.89)
  Week 25 Day 1,n=0,0,1,0,0,1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  Week 25 Day 1,n=0,0,1,0,0,1 |  |  | 0.0 (NA) — Standard deviation could not be calculated for single participant. |  |  | -8.3 (NA) — Standard deviation could not be calculated for single participant.
  Week 29 Day 1,n=0,0,0,0,0,2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2
  Week 29 Day 1,n=0,0,0,0,0,2 |  |  |  |  |  | -8.3 (11.79)
  Week 33 Day 1,n=0,0,1,0,1,2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 2
  Week 33 Day 1,n=0,0,1,0,1,2 |  |  | 8.3 (NA) — Standard deviation could not be calculated for single participant. |  | 0.0 (NA) — Standard deviation could not be calculated for single participant. | -8.3 (11.79)
  Week 37 Day 1,n=0,0,1,0,0,3: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 3
  Week 37 Day 1,n=0,0,1,0,0,3 |  |  | 0.0 (NA) — Standard deviation could not be calculated for single participant. |  |  | -2.8 (4.81)
  Week 41 Day 1,n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Week 41 Day 1,n=0,0,1,0,0,0 |  |  | 8.3 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Week 45 Day 1,n=0,0,1,0,0,1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  Week 45 Day 1,n=0,0,1,0,0,1 |  |  | -8.3 (NA) — Standard deviation could not be calculated for single participant. |  |  | 0.0 (NA) — Standard deviation could not be calculated for single participant.
  Week 49 Day 1,n=0,0,1,0,0,2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 2
  Week 49 Day 1,n=0,0,1,0,0,2 |  |  | 16.7 (NA) — Standard deviation could not be calculated for single participant. |  |  | -8.3 (0.00)
  Week 61 Day 1,n=0,0,1,0,0,1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  Week 61 Day 1,n=0,0,1,0,0,1 |  |  | 16.7 (NA) — Standard deviation could not be calculated for single participant. |  |  | -16.7 (NA) — Standard deviation could not be calculated for single participant.

26. Secondary Outcome: Change From Baseline in Brief Pain Inventory - Short Form (BPI-SF): Pain Intensity- Pain at Worst in Last 24 Hours
Description: BPI-SF is 9-item self-administered questionnaire. Pain intensity score was calculated from the four items (items 3, 4, 5 and 6) for worst pain, least pain, average pain and current pain. Worst pain in last 24 hours was rated from 0 (no pain) to 10 (pain as bad as you can imagine). Baseline is defined as the latest non-missing assessment time-point prior to the first study treatment dose (latest up to Week 1 Day 1). Change from Baseline was calculated as post-Baseline visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Week 1 Day 1) and on Day 1 of Weeks 2, 3, 4, 5, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 61, 73, 85, 97
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 9 | 5 | 4 | 10 | 19 | 17
Scores on a scale
  Week 2 Day 1,n=9,5,4,9,14,13: number analyzed (Participants) | 9 | 5 | 4 | 9 | 14 | 13
  Week 2 Day 1,n=9,5,4,9,14,13 | 0.1 (2.62) | 0.8 (2.86) | -2.3 (1.71) | 0.0 (1.12) | 0.0 (2.91) | 0.2 (1.48)
  Week 3 Day 1,n=8,3,4,10,16,15: number analyzed (Participants) | 8 | 3 | 4 | 10 | 16 | 15
  Week 3 Day 1,n=8,3,4,10,16,15 | 0.5 (1.77) | -1.7 (1.53) | -1.8 (1.89) | -1.0 (2.05) | 0.3 (3.26) | 0.0 (1.51)
  Week 4 Day 1,n=8,4,3,8,16,15: number analyzed (Participants) | 8 | 4 | 3 | 8 | 16 | 15
  Week 4 Day 1,n=8,4,3,8,16,15 | 0.4 (1.92) | 0.5 (1.91) | -1.3 (1.15) | -0.8 (1.28) | 0.2 (2.81) | 0.4 (1.76)
  Week 5 Day 1,n=6,4,4,10,19,17: number analyzed (Participants) | 6 | 4 | 4 | 10 | 19 | 17
  Week 5 Day 1,n=6,4,4,10,19,17 | -0.8 (3.06) | -0.3 (1.26) | -1.0 (0.82) | -0.9 (2.13) | 0.7 (3.38) | -0.2 (1.78)
  Week 9 Day 1,n=3,4,3,8,10,13: number analyzed (Participants) | 3 | 4 | 3 | 8 | 10 | 13
  Week 9 Day 1,n=3,4,3,8,10,13 | 1.3 (1.53) | 1.3 (0.96) | -0.3 (2.52) | -0.5 (2.07) | 0.2 (2.49) | -0.4 (2.40)
  Week 13 Day 1,n=2,3,1,5,7,7: number analyzed (Participants) | 2 | 3 | 1 | 5 | 7 | 7
  Week 13 Day 1,n=2,3,1,5,7,7 | 0.5 (0.71) | 2.0 (3.00) | 2.0 (NA) — Standard deviation could not be calculated for single participant. | 0.2 (1.92) | -1.7 (2.21) | -0.4 (2.15)
  Week 17 Day 1,n=2,4,2,5,3,8: number analyzed (Participants) | 2 | 4 | 2 | 5 | 3 | 8
  Week 17 Day 1,n=2,4,2,5,3,8 | 2.5 (7.78) | 3.5 (4.36) | -0.5 (4.95) | -0.8 (3.11) | -1.3 (1.15) | -0.5 (2.20)
  Week 21 Day 1,n=1,2,2,5,3,6: number analyzed (Participants) | 1 | 2 | 2 | 5 | 3 | 6
  Week 21 Day 1,n=1,2,2,5,3,6 | 2.0 (NA) — Standard deviation could not be calculated for single participant. | 0.5 (0.71) | -2.5 (0.71) | -0.2 (2.49) | -2.3 (4.04) | 1.0 (1.79)
  Week 25 Day 1,n=0,0,1,2,3,4: number analyzed (Participants) | 0 | 0 | 1 | 2 | 3 | 4
  Week 25 Day 1,n=0,0,1,2,3,4 |  |  | 3.0 (NA) — Standard deviation could not be calculated for single participant. | 0.0 (0.00) | -1.3 (5.69) | -1.0 (1.15)
  Week 29 Day 1,n=0,0,1,3,2,4: number analyzed (Participants) | 0 | 0 | 1 | 3 | 2 | 4
  Week 29 Day 1,n=0,0,1,3,2,4 |  |  | -3.0 (NA) — Standard deviation could not be calculated for single participant. | -0.7 (1.15) | -3.5 (0.71) | 0.8 (4.19)
  Week 33 Day 1,n=0,0,1,3,2,2: number analyzed (Participants) | 0 | 0 | 1 | 3 | 2 | 2
  Week 33 Day 1,n=0,0,1,3,2,2 |  |  | 1.0 (NA) — Standard deviation could not be calculated for single participant. | 0.7 (1.15) | -1.5 (2.12) | -1.0 (1.41)
  Week 37 Day 1,n=0,0,1,3,0,4: number analyzed (Participants) | 0 | 0 | 1 | 3 | 0 | 4
  Week 37 Day 1,n=0,0,1,3,0,4 |  |  | 0.0 (NA) — Standard deviation could not be calculated for single participant. | 1.7 (2.08) |  | 0.0 (1.41)
  Week 41 Day 1,n=0,0,1,3,1,1: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1 | 1
  Week 41 Day 1,n=0,0,1,3,1,1 |  |  | -1.0 (NA) — Standard deviation could not be calculated for single participant. | 1.3 (1.53) | -3.0 (NA) — Standard deviation could not be calculated for single participant. | -1.0 (NA) — Standard deviation could not be calculated for single participant.
  Week 45 Day 1,n=0,0,1,2,1,3: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 3
  Week 45 Day 1,n=0,0,1,2,1,3 |  |  | 1.0 (NA) — Standard deviation could not be calculated for single participant. | 2.5 (2.12) | -1.0 (NA) — Standard deviation could not be calculated for single participant. | 1.7 (1.15)
  Week 49 Day 1,n=0,0,1,3,1,3: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1 | 3
  Week 49 Day 1,n=0,0,1,3,1,3 |  |  | 2.0 (NA) — Standard deviation could not be calculated for single participant. | 0.3 (1.53) | -3.0 (NA) — Standard deviation could not be calculated for single participant. | 2.7 (2.52)
  Week 61 Day 1,n=0,0,1,1,1,1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 1
  Week 61 Day 1,n=0,0,1,1,1,1 |  |  | -2.0 (NA) — Standard deviation could not be calculated for single participant. | 0.0 (NA) — Standard deviation could not be calculated for single participant. | -3.0 (NA) — Standard deviation could not be calculated for single participant. | 3.0 (NA) — Standard deviation could not be calculated for single participant.
  Week 73 Day 1,n=0,0,0,1,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 0
  Week 73 Day 1,n=0,0,0,1,1,0 |  |  |  | 0.0 (NA) — Standard deviation could not be calculated for single participant. | -2.0 (NA) — Standard deviation could not be calculated for single participant. |
  Week 85 Day 1,n=0,0,0,1,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 0
  Week 85 Day 1,n=0,0,0,1,1,0 |  |  |  | 3.0 (NA) — Standard deviation could not be calculated for single participant. | -3.0 (NA) — Standard deviation could not be calculated for single participant. |
  Week 97 Day 1,n=0,0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Week 97 Day 1,n=0,0,0,0,1,0 |  |  |  |  | -3.0 (NA) — Standard deviation could not be calculated for single participant. |

27. Other Pre Specified Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs) Until End of the Study
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, any other situation according to medical or scientific judgement, or is associated with liver injury and impaired liver function. Number of Participants With any AEs and SAEs collected from start of the treatment until end of the study were reported.
Time Frame: Up to 3 years and 11 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21
Participants
  Any AEs | 10 | 6 | 4 | 10 | 22 | 21
  Any SAEs | 4 | 2 | 0 | 1 | 6 | 7

28. Other Pre Specified Outcome: Number of Participants With AEs Leading to Any Dose Reduction or Delays Until End of the Study
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of Participants with AEs leading to any dose reduction or delays from start of the treatment until end of the study were reported.
Time Frame: Up to 3 years and 11 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21
Participants
  Dose reduction | 4 | 1 | 0 | 7 | 10 | 7
  Dose delay | 5 | 2 | 4 | 8 | 15 | 12

29. Other Pre Specified Outcome: Number of Participants Who Withdrew Due to Toxicity and Changes in Safety Assessment Until End of the Study
Description: Number of participants who withdrew due to toxicity and changes in safety assessment including laboratory parameters and vital signs from start of the treatment until end of the study were reported.
Time Frame: Up to 3 years and 11 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
Number analyzed (Participants) | 10 | 6 | 4 | 10 | 22 | 21
Participants | 6 | 2 | 2 | 3 | 8 | 4

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected up to 3 years and 11 months
Description: All-cause mortality, non-SAES and SAEs were assessed using All Treated Population which consisted of all participants who received at least one dose of GSK525762 or abiraterone or enzalutamide.
Arm/Group | GSK525762 60 mg+Abiraterone 1000 mg | GSK525762 60 mg Alternate+Abiraterone 1000 mg | GSK525762 40 mg+Abiraterone 1000 mg | GSK525762 80 mg+Enzalutamide 160 mg | GSK525762 60 mg+Enzalutamide 160 mg | GSK525762 60 mg Alternate+Enzalutamide 160 mg
All-Cause Mortality (participants affected / at risk) | 9/10 | 2/6 | 2/4 | 7/10 | 8/22 | 10/21
Serious Adverse Events (participants affected / at risk) | 4/10 | 2/6 | 0/4 | 1/10 | 6/22 | 7/21
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6 | 4/4 | 10/10 | 22/22 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK525762 60 mg+Abiraterone 1000 mg (N=10) | GSK525762 60 mg Alternate+Abiraterone 1000 mg (N=6) | GSK525762 40 mg+Abiraterone 1000 mg (N=4) | GSK525762 80 mg+Enzalutamide 160 mg (N=10) | GSK525762 60 mg+Enzalutamide 160 mg (N=22) | GSK525762 60 mg Alternate+Enzalutamide 160 mg (N=21)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK525762 60 mg+Abiraterone 1000 mg (N=10) | GSK525762 60 mg Alternate+Abiraterone 1000 mg (N=6) | GSK525762 40 mg+Abiraterone 1000 mg (N=4) | GSK525762 80 mg+Enzalutamide 160 mg (N=10) | GSK525762 60 mg+Enzalutamide 160 mg (N=22) | GSK525762 60 mg Alternate+Enzalutamide 160 mg (N=21)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 4 (6) | 4 (6) | 9 (15) | 13 (15)
Nausea (Gastrointestinal disorders) | 7 (9) | 3 (3) | 1 (2) | 6 (7) | 8 (9) | 11 (17)
Fatigue (General disorders) | 7 (8) | 2 (2) | 0 (0) | 3 (3) | 11 (18) | 7 (9)
Dysgeusia (Nervous system disorders) | 5 (7) | 2 (2) | 2 (3) | 2 (5) | 7 (11) | 10 (11)
Asthenia (General disorders) | 0 (0) | 3 (4) | 4 (5) | 2 (7) | 8 (11) | 11 (14)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (5) | 2 (3) | 6 (10) | 7 (10)
Vomiting (Gastrointestinal disorders) | 5 (6) | 1 (1) | 0 (0) | 2 (2) | 6 (11) | 7 (10)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0) | 3 (4) | 7 (8) | 3 (3)
Platelet count decreased (Investigations) | 4 (6) | 2 (5) | 1 (1) | 4 (17) | 4 (5) | 4 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 9 (14) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 6 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 3 (4) | 0 (0) | 4 (5) | 0 (0) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 4 (5)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 3 (3) | 3 (4)
Amylase increased (Investigations) | 3 (3) | 0 (0) | 2 (3) | 2 (3) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 3 (4) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 2 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT03150056/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT03150056/SAP_001.pdf